CLINICAL TRIAL: NCT05867602
Title: Clinical Efficacy of High-dose Albumin Administration Versus Standard Dose in Patients With Advanced Cirrhosis: Open Label Randomized Clinical Trial
Brief Title: High Dose Albumin in Refractory Ascites
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Prasun Kumar Jalal, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-49043
Record Dates: First submitted 2023-04-20; First posted 2023-05-22 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Ascites
Keywords: refractory ascites; liver cirrhosis; HRS; High dose albumin
MeSH Terms: conditions — Ascites; Liver Cirrhosis | interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): the intervention group will receive intravenous human albumin at a dose of (1g/kg), with a minimum dose of 50g and a maximum dose of 100g, plus SOC
  Interventions: Drug: Albumin
- Control arm (No Intervention): the control arm will receive the standard of care (SOC), including moderate sodium restriction, maximal daily tolerated doses of diuretics, and post-paracentesis albumin

INTERVENTIONS:
Drug: Albumin — intravenous human albumin at a dose of (1g/kg), with a minimum dose of 50g and a maximum dose of 100g
  Other Names: High dose albumin (HA)
  Arms: Intervention arm

SUMMARY:
Advanced cirrhosis with complications is a serious problem imposing a heavy financial burden on health care system. Moreover, ascites is associated with increase in mortality rates among cirrhotic patients. Ascites pathogenesis is multifactorial including: portal hypertension; splanchnic and peripheral arterial vasodilation; and neurohumoral activation. Current management strategies include dietary sodium restriction and diuretic therapy, however, this strategy put patients at the risk of intravascular volume depletion, renal impairment, hepatic encephalopathy and hyponatremia. Moreover, around 10% of patients do not respond to this strategy (termed: diuretics resistant) with 50% of them die within 6 months. This sub-group is managed by frequent large volume paracentesis along with intravenous albumin administration and are usually considered for liver transplantation (LT) and TIPS. Nonetheless, Frequent paracentesis increases the risk of infection, bleeding, bowel perforation, paracentesis-induced circulatory dysfunction (PICD) and renal dysfunction in this sub-group of patients. The beneficial effect of human albumin might result from blood volume expansion tapering activated vasoconstrictor and sodium-retaining systems improving renal perfusion, hence regular infusion of albumin may be beneficial to prevent development of ascites and to improve survival. The positive effects of albumin are supported by previous studies; Romanelli et al, showed a significant increase in survival rate among cirrhotic patients with ascites when compared to those who did not receive albumin. Moreover, a randomized multicenter open label trial published in lancet last year, demonstrated that long term albumin administration improved 18-month survival, decreased the use of paracentesis and decrease in the incidence of cirrhosis related complications among cirrhotic patients with ascites. As of today, there's a limited use of regular high dose albumin in cirrhotic patients with ascites in US, despite being used elsewhere in the world as previously stated.

The investigators wish to study long-term efficacy of human albumin administration in patients with decompensated cirrhosis to assess safety and efficacy, and prevention of complications of cirrhosis.

DETAILED DESCRIPTION:
Patients with advanced liver disease often has low serum albumin level. The Infusion of human albumin is a standard of care after removal of ascitic fluid in patients with cirrhosis with refractory ascites. The objective of the study is to prove that regular infusion of albumin prevents formation of fluid in abdomen (ascites) or pleural fluid (Hydrothorax) and thus reduces the requirement of paracentesis or thoracentesis, and prevent complications.

The Primary endpoints are: (1) Number of paracentesis/thoracentesis needed and volume of fluid removed per month and if there is any reduction in frequency or volume after high-dose albumin administration; (2) Twelve-month mortality or transplant. Secondary endpoints are: (1) Improvement of MELD score; (2) Cumulative diuretic dosage; (3) Development of hyponatremia or hyperkalemia as potential diuretic-induced side-effects; (4) Incidence of cirrhosis related complications (spontaneous bacterial peritonitis, other bacterial infections, renal impairment, hepatorenal syndrome, hepatic encephalopathy and gastrointestinal bleeding related to portal hypertension); (5) Quality of life; (6) Number and duration of hospital admissions; and (7) Treatment cost-effectiveness.

The research design is a prospective, parallel, randomized, open label clinical trial. The target trial population comprises of patients with advanced cirrhosis. Eligible patients will be randomized into either one of two categories: 1) the control group will receive the standard of care (SOC) including moderate sodium restriction and maximal daily tolerated doses of diuretics, and 2) the Intervention group will receive intravenous human albumin at a dose (1g/kg, with minimum dose of 50g and maximum dose of 100g) weekly plus SOC.

In both groups, when large-volume paracentesis is needed, the patient will receive human albumin in the dose of 6-8 g/L of ascites removed as SOC.

Inclusion Criteria:

1. Age > 18 years.
2. patients diagnosed with liver cirrhosis. Refractory ascites which is defined as ascites failing to resolve after maximum tolerable dose of diuretics, and usually require frequent paracentesis.

Exclusion Criteria:

1. Patients < 18y and patients with no history of liver cirrhosis
2. patients with refractory ascites but have trans-jagular intrahepatic portosystemic shunts (TIPS) with previous 3 months
3. Patients with ascites due to other causes, including cardiac, malignant Procedure Eligible patients will be identified by the PI and the research team. Participants will be approached to participate in the study. The research coordinator will fully explain the study procedures, and if the patient is willing to participate, he or she will sign the informed consent. After signing the informed consent, eligible patients will be randomly assigned into two groups: 1) the control arm will receive the standard of care (SOC), including moderate sodium restriction, maximal daily tolerated doses of diuretics, and post-paracentesis albumin, and 2) the intervention group will receive intravenous human albumin at a dose of (1g/kg), with a minimum dose of 50g and a maximum dose of 100g, plus SOC. patients will be randomly assigned (1:1) to either of these two groups.

In both groups, when large-volume paracentesis is needed, the participant will receive human albumin in the dose of 6-8 g/L of ascites removed.

No concomitant medications are withheld during the study. After enrollment, participants will be assessed by a physician monthly for up to one year or study interruption or liver transplant or death. In both groups with refractory ascites, most of the patient require weekly or biweekly monitoring and paracentesis. The investigators plan to approach the patients during these visits to get the consent and administer the extra albumin dose.

In each visit, ascites severity will be evaluated with hemodynamic status, weight, new symptoms, and diuretic dose. Each visit may last 15 minutes or more.

Patients who consent to the study will complete a self-administered questionnaire to assess health-related quality of life (using CLDQ, CLDQ-HCV and CLDQ- NASH Questionnaires). Each patient response will be coded to ensure privacy, and the coded data will be entered into a collection sheet with no protected health information (PHI) gathered during the survey. The investigators will give the questionnaire: at the time of enrollment and at the 6 and 12 month time points

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. patients diagnosed with liver cirrhosis.
3. Refractory ascites which is defined as ascites failing to resolve after maximum tolerable dose of diuretics, and usually require frequent paracentesis.

Exclusion Criteria:

1. Patients < 18y
2. patients with no history of liver cirrhosis
3. patients with refractory ascites but have transjagular intrahepatic portosystemic shunts (TIPS) with previous 3 months
4. Patients with ascites due to other causes, including cardiac, malignant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Number of large volume paracentesis needed | 1 year
  Number of paracentesis/thoracentesis needed.
The volume of fluid removed in liters per after high-dose albumin administration | 1 year
  Measuring the fluid amount removed each paracentesis and compare it to before High dose albumin administration

SECONDARY OUTCOMES:
Incidence of cirrhosis related complications (spontaneous bacterial peritonitis, other bacterial infections, renal impairment, hepatorenal syndrome, hepatic encephalopathy and gastrointestinal bleeding related to portal hypertension). | 1 year
  Each attack of decompensation will be documented during enrollment. We will compare number of decompensation episodes in each group
Diuretics dosage assessment | 1 Year
  Trend for Dosage of diuretics required in mg during the enrollment period.
Liver related quality of life assessment. | 1 year
  Liver related quality of life assessment.
Mortality at 1 year after enrollment | 1 year
  Twelve-month mortality
Number and duration of hospital admissions | 1 year
  Number of visits to ER, hospital admissions will also be assessed
Treatment cost-effectiveness. | 1year
  Cost of albumin vs cost of paracentesis and paracentesis related hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Prasun Jalal, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor St' Lukes Medical center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Pascoli M, Ceranto E, De Nardi P, Donato D, Gatta A, Angeli P, Pontisso P. Hospitalizations Due to Cirrhosis: Clinical Aspects in a Large Cohort of Italian Patients and Cost Analysis Report. Dig Dis. 2017;35(5):433-438. doi: 10.1159/000458722. Epub 2017 Mar 1. PMID 28245467
- [Background] Gines P, Quintero E, Arroyo V, Teres J, Bruguera M, Rimola A, Caballeria J, Rodes J, Rozman C. Compensated cirrhosis: natural history and prognostic factors. Hepatology. 1987 Jan-Feb;7(1):122-8. doi: 10.1002/hep.1840070124. PMID 3804191
- [Background] Schmidt ML, Barritt AS, Orman ES, Hayashi PH. Decreasing mortality among patients hospitalized with cirrhosis in the United States from 2002 through 2010. Gastroenterology. 2015 May;148(5):967-977.e2. doi: 10.1053/j.gastro.2015.01.032. Epub 2015 Jan 23. PMID 25623044
- [Background] Pedersen JS, Bendtsen F, Moller S. Management of cirrhotic ascites. Ther Adv Chronic Dis. 2015 May;6(3):124-37. doi: 10.1177/2040622315580069. PMID 25954497
- [Background] Moore KP, Aithal GP. Guidelines on the management of ascites in cirrhosis. Gut. 2006 Oct;55 Suppl 6(Suppl 6):vi1-12. doi: 10.1136/gut.2006.099580. No abstract available. PMID 16966752
- [Background] Pache I, Bilodeau M. Severe haemorrhage following abdominal paracentesis for ascites in patients with liver disease. Aliment Pharmacol Ther. 2005 Mar 1;21(5):525-9. doi: 10.1111/j.1365-2036.2005.02387.x. PMID 15740535
- [Background] Romanelli RG, La Villa G, Barletta G, Vizzutti F, Lanini F, Arena U, Boddi V, Tarquini R, Pantaleo P, Gentilini P, Laffi G. Long-term albumin infusion improves survival in patients with cirrhosis and ascites: an unblinded randomized trial. World J Gastroenterol. 2006 Mar 7;12(9):1403-7. doi: 10.3748/wjg.v12.i9.1403. PMID 16552809